CLINICAL TRIAL: NCT04866459
Title: MYO-SHARE: MYO-MRI in Neuromuscular Diseases
Acronym: MYO-SHARE
Status: Enrolling by invitation | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MYO-SHARE
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuromuscular Diseases (NMDs) affect > 7 million people worldwide. NMDs are often difficult to accurately diagnose, with over 200 different genetic causes with overlapping clinical presentations. Muscle Magnetic Resonance Imaging (Muscle MRI) allows for non-invasive, comprehensive, and reproducible evaluation of disease-affected and spared muscles. The selective replacement of muscle tissue by fat is the main contributor to pathological patterns determined by T1-weighted Muscle MRI. Although the diagnostic utility of Muscle MRI has been emphasized in the last years, the very low incidence of NMDs (rate .01 to 15 per 100,000 population), and the challenge to attain sufficient sample sizes to study the imaging characteristics of these patients have limited their acceptance as first-line, non-invasive diagnostic procedures. The purpose of this study is to examine the selective pattern of muscle pathology as detected by MRI of different sub-types of NMDs and validate this technique as an important and helpful non-invasive diagnostic screening tool.

This study will prospectively assemble a well-defined cohort of 1000 patients with NMDs undergoing whole body Muscle MRI from 7 Canadian and 7 international centers. It will develop a high-standard methodological approach for MRI diagnosis in this cohort, based on T1 weighted imaging characteristics, and will validate this method by testing the developed algorithm in a different cohort of patients. Muscle MRI scans will be collected by a well-established network of neuromuscular disease (NMD) centers to ensure comparability between the different centers.

DETAILED DESCRIPTION:
The primary objectives of this study are:

1. Establish a large, well-defined international cohort of patients with NMDs with Muscle MRI
2. Identify diagnostic patterns of muscle involvement for patients with rare NMDs using Muscle MRI
3. Validate diagnostic patterns of muscle pathology detected by MRI for patients with rare NMDs

Additional objective of this study:

1. Provide practice-changing information regarding the optimal use of Muscle MRI in patients suspected of having an NMD

Whole Body Muscle MRI is emerging as a tool to identify diseased muscles that are not readily evaluated by clinical examination, where patterns of involvement may be associated with specific Neuromuscular Diseases (NMDs) and may provide additional evidence to rule in/out a particular genetic variant. Previous studies have outlined more common NMDs, and the majority of rare NMDs do not have large cohorts of patients to clearly establish "specific" muscle patterns. Progress has also been limited by a lack of international standards to acquire MRIs and identifying MRI patterns of affected muscles.

By collectively pooling MRI scans for patients with different NMDs, this study will help improve the characterization of selective patterns of muscle atrophy, fatty degeneration, and muscle edema in specific diseases and avoid misdiagnosis of genetic or acquired NMDs. Recognizing patterns of pathology by muscle or nerve imaging can help to guide or confirm genetic testing and to avoid the more invasive procedure of a muscle biopsy. Finally, this project will inform quantitative MRI approaches by identifying the most appropriate regions of interest to be scanned in clinical trials for specific NMDs.

ELIGIBILITY:
Inclusion Criteria:

1.Clinical diagnosis of neuromuscular disease: Potential participants will have a diagnosis of NMD, based on clinical testing, electrodiagnostic studies and antibody testing or genetic testing of a pathogenic variant based on the American College of Medical Genetics criteria [63]. Standard-of-care assessments include a detailed NMD examination by neurogenetics or neuromuscular physician, a three-generation family history, genetic testing, electrophysiological studies, and standard myopathy serology (e.g., creatine kinase level), muscle biopsy, muscle ultrasound, etc. will be considered for this study.

Exclusion Criteria:

1. Patients with contraindications to MRI 1.1 Including non-MR compatible cardiac pacemaker or electronic devices 1.2 Severe claustrophobia
2. Patients with clinical presentation not consistent with confirmed NMD
3. Patients with advanced disease with severe quadriparesis (Medical Research Council Muscle Rating score of <3 in >10 muscle groups) or asymptomatic patients, as severe fatty replacement of muscle tissue in the late disease of most muscles or normal scans, will limit the value of diagnosis by imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuromuscular Diseases
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2031-05-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
1. Provide a very large and unique, well-defined international cohort of genetically diagnosed patients with NMDs and whole-body Muscle MRI scans with carefully curated phenotypes | 10 years
  This study will provide a very large and unique, well-defined international cohort (1000 participants) of genetically diagnosed patients with NMDs and whole-body Muscle MRI scans with carefully curated phenotypes. This study aims to provide the diagnostic rate of Muscle MRI in a well-defined cohort and assess the diagnostic value of certain selective patterns of pathology obtained by T1 weighted Muscle MRI.
2. Characterize disease progression and affected muscle regions of interest | 10 years
  Although diagnostic muscle MRI is resulting in an increased pooling of MRI data, often these data are never published/publicly shared and are lost to science. Combining these data through effective networking with MYO-Share will help further define the spectrum of selective patterns of pathology (including muscles not normally biopsied, e.g. diaphragm, trunk, neck and head), to detect patterns that may suggest a common underlying mechanism or pathway. This study will also help characterize disease progression and affected muscle regions of interest for targeted biopsies and relevant for quantitative MRI.
3. Provide the diagnostic rate of Muscle MRI in a well-defined cohort and assess the diagnostic value of certain selective patterns of pathology obtained by T1 weighted Muscle MRI | 10 years
  In order to extend both the acquisition of imaging data and the expertise in data analysis and pattern recognition, it will be important to clearly demonstrate the added diagnostic value. If Muscle MRI is demonstrated to have a high diagnostic accuracy, this would benefit patients as it could confirm a genetic diagnosis and avoid unnecessary muscle biopsies.

SECONDARY OUTCOMES:
1. Provide practice-changing information regarding the optimal use of Muscle MRI in patients suspected of having a NMD | 10 years
  This study will provide practice-changing information regarding the optimal use of Muscle MRI in patients suspected of having a NMD, impacting both patients as well as the healthcare system that cares for them. This current study will serve as a proof-of-principle of the effectiveness of MYO-Share and demonstrate potential to study larger clinical and research cohorts of both pediatric and adult patients with NMD. To increase awareness and stimulate further research into this area of diagnostic care, we will present our findings at national and international conferences and publish our findings in a high impact peer reviewed journals. Presentations will also be delivered at patient-driven community events.

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Warman, MD, PhD, Principal Investigator — The Ottawa Hospital, University of Ottawa, Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No